CLINICAL TRIAL: NCT01088490
Title: Hydrogen Sulfide as Prognostic Factor
Acronym: H2S-1
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Podbregar Matej, Prof., University Medical Centre Ljubljana
Other Study IDs: H2S_1
Record Dates: First submitted 2010-03-12; First posted 2010-03-17 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Mortality; Shock
Keywords: Hydrogen sulfide; critically ill; mortality
MeSH Terms: conditions — Shock; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- critically ill: Critically ill patients admitted to ICU

SUMMARY:
Hydrogen sulfide (H2S), better known as a poisonous gas, has emerged as the third gaseous transmitter in mammals, next to nitric oxide (NO) and carbon monoxide (CO). Increased production and higher serum concentrations were shown in inflammatory diseases, septic shock and stroke. The investigators will test the hypothesis that higher serum H2S concentrations on admission to intensive care unit (ICU) are linked with higher mortality in patients with shock of any reason.

DETAILED DESCRIPTION:
Hydrogen sulfide (H2S), better known as a poisonous gas, has lately emerging as a third gaseous transmitter in mammals, next to nitric oxide (NO) and carbon monoxide (CO). H2S is present in most human tissues in concentrations up to 50 μM. Most of it is synthesized in brain, cardiovascular system, kidneys and liver. In human tissues H2S is synthesized from L-cysteine by two enzymes cystathionine-γ-lyase and cystathionine-β-synthase. H2S works by stimulating ATP sensitive potassium channels and is involved in regulation of vascular tone, myocardial contractility, insulin secretion and neurotransmission. In numerous animal models, H2S deficiency was shown in arterial and pulmonary arterial hypertension, Alzheimer's disease and liver cirrhosis. Increased production and higher serum concentrations were shown in inflammatory diseases, septic shock and stroke.

Most of studies so far were conducted on animals and already show some therapeutic potentials. In available literature there have been no studies in humans focused on H2S concentrations in critically ill and its prognostic value.

Hypothesis We will test the hypothesis that higher serum H2S concentrations on admission to ICU are linked with higher mortality in patients with shock of any reason.

Serum H2S concentrations are related to treatment support with vaso-active drugs (noradrenalin, epinephrine).

Material and methods In the study we will include adult patients admitted to medical ICU due to shock of any reason. Shock is defined as systemic arterial pressure lower than 90mmHg or drop for systemic arterial pressure at least 40mmHg for 15minutes or more with elevation of serum lactate value.

Patients will be included on basis of clinical appearance of shock - hypotension or need for vasopressors, brady- or tachycardia, signs of peripheral hypo perfusion, oliguria and changes in mental status.

Exclusion criteria: patient younger then 18years and patients not in shock

From blood samples drawn on admission to ICU we will measure H2S concentration. H2S concentration will be measured spectrophotometrically5 as first described in 19496 and further refined in 19657. Spectrophotometrical determination of H2S concentration in tissue and plasma was previously used by many researchers.3,8-11 Blood samples will be centrifuged as quickly after collection to obtain plasma. 200 μL of plasma will be mixed with pre-prepared solution of 100 μL 10% (wt/vol) trichloroacetic acid and 60 μL 1% (wt/vol) zinc acetate, to trap dissolved H2S. The mixture will be frozen at 20 C until further analysis.

After sufficient number of samples will be obtained, we will measure H2S concentration in series. 40µL 20 µM N,N-dimethyl-p-phenylenediamine sulfate in 7,2 M HCl and 40µL 30 µM FeCl3 v 1,2 M HCl will be added to unfrozen samples. After 10-20 min incubation at room temperature final mixtures will be centrifuged at 9000 rpm for 5 minutes to remove precipitate. After centrifugation absorption at 670 nm will be measured with spectrophotometer. All analysis will be done in duplicates.

Calibration curve of absorbance versus sulfide concentration will be obtained from known concentration of Na2S (0,699 µM - 69,93 µM) and concentrations of H2S in plasma calculated.

Impact of plasma H2S concentration on admission to ICU on ICU mortality will be observed trough nonparametric statistical analysis.

Expectations We hypothesize that higher serum H2S concentrations on admission to ICU in patients with shock of any cause are indicators of severity of shock and cardiovascular deterioration, related to treatment support with vaso-active drugs (noradrenalin, epinephrine). Thus higher serum H2S concentrations are expected to be better prognostic factor of ICU mortality in patients with shock than currently established lactic acid.

ELIGIBILITY:
Inclusion Criteria:

* shock ( systemic arterial pressure less then 120mmHg, elevated lactate > 2.5mmol/L)

Exclusion Criteria:

* patients admitted due to intoxication with H2S

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients how are admitted in shock or hemodynamicaly unstable ino intensive care
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Prognostic value of H2S | In hospital; ICU mortality 30days
  relationship between H2S and mortality of patients during intensive care treatment,
  comparison of H2S and lactate prognostic value

SECONDARY OUTCOMES:
Correlation of H2S with vasopressor requirements | ICU treatmennt 30days
  relationship between H2S and dose of vasopressors (noradrenaline, epinephrine) used

CONTACTS AND LOCATIONS:
Overall Officials: Matej Podbregar, MD PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Center, Ljubljana, Slovenia, Slovenia

REFERENCES:
- [Background] Lowicka E, Beltowski J. Hydrogen sulfide (H2S) - the third gas of interest for pharmacologists. Pharmacol Rep. 2007 Jan-Feb;59(1):4-24. PMID 17377202
- [Background] Hui Y, Du J, Tang C, Bin G, Jiang H. Changes in arterial hydrogen sulfide (H(2)S) content during septic shock and endotoxin shock in rats. J Infect. 2003 Aug;47(2):155-60. doi: 10.1016/s0163-4453(03)00043-4. PMID 12860150
- [Background] Mok YY, Atan MS, Yoke Ping C, Zhong Jing W, Bhatia M, Moochhala S, Moore PK. Role of hydrogen sulphide in haemorrhagic shock in the rat: protective effect of inhibitors of hydrogen sulphide biosynthesis. Br J Pharmacol. 2004 Dec;143(7):881-9. doi: 10.1038/sj.bjp.0706014. Epub 2004 Oct 25. PMID 15504752
- [Background] Li L, Bhatia M, Zhu YZ, Zhu YC, Ramnath RD, Wang ZJ, Anuar FB, Whiteman M, Salto-Tellez M, Moore PK. Hydrogen sulfide is a novel mediator of lipopolysaccharide-induced inflammation in the mouse. FASEB J. 2005 Jul;19(9):1196-8. doi: 10.1096/fj.04-3583fje. Epub 2005 Apr 29. PMID 15863703
- [Background] Lawrence NS, Davis J, Compton RG. Analytical strategies for the detection of sulfide: a review. Talanta. 2000 Aug 16;52(5):771-84. doi: 10.1016/s0039-9140(00)00421-5. PMID 18968036
- [Background] Zhang H, Zhi L, Moore PK, Bhatia M. Role of hydrogen sulfide in cecal ligation and puncture-induced sepsis in the mouse. Am J Physiol Lung Cell Mol Physiol. 2006 Jun;290(6):L1193-201. doi: 10.1152/ajplung.00489.2005. Epub 2006 Jan 20. PMID 16428267
- [Background] Collin M, Thiemermann C. Hydrogen sulfide and sulfite: novel mediators in the pathophysiology of shock and inflammation. Shock. 2005 Dec;24(6):595-6. doi: 10.1097/01.shk.0000188328.59770.25. No abstract available. PMID 16317393
- [Background] Abe K, Kimura H. The possible role of hydrogen sulfide as an endogenous neuromodulator. J Neurosci. 1996 Feb 1;16(3):1066-71. doi: 10.1523/JNEUROSCI.16-03-01066.1996. PMID 8558235
- [Derived] Goslar T, Mars T, Podbregar M. Total plasma sulfide as a marker of shock severity in nonsurgical adult patients. Shock. 2011 Oct;36(4):350-5. doi: 10.1097/SHK.0b013e31822bcfd0. PMID 21897337